CLINICAL TRIAL: NCT05678231
Title: Use of the Disposable Zero Degree Knee Postoperative Positioner for Improved Early Knee Extension and Self-Reported Outcomes Following Total Knee Arthroplasty
Brief Title: Zero Degree Knee Positioner for Improved Earley Knee Extension Following Total Knee Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Midlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1983229
Record Dates: First submitted 2022-12-13; First posted 2023-01-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee arthroplasty; Osteoarthritis; Total knee replacement
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Patients electing to undergo primary TKA will be recruited into the study and randomized to receive and follow the ZDK protocol post-operatively or standard of care rehabilitation instructions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patients will receive standard of care instructions rehabilitation instructions following total knee replacement.
- Zero Degree Knee (Experimental): Patients will receive the Zero Degree Knee device and instructions for use following total knee replacement.
  Interventions: Device: Zero Degree Knee Positioner

INTERVENTIONS:
Device: Zero Degree Knee Positioner — The Zero Degree Knee (ZDK) positioning device is a knee extension pillow designed to simplify knee extension exercise following TKA surgery.
  Arms: Zero Degree Knee

SUMMARY:
Studies have demonstrated that early rehabilitation interventions following knee arthroplasty (TKA) can shorten the time needed to regain baseline extension/full extension and gait mechanics. As telehealth visits and home-based rehabilitation increases with advancements in technology, much of this rehabilitation is projected to be performed at home. The purpose of this study is to prospectively evaluate early post-operative knee extension and self-reported outcomes in patients using the Zero Degree Knee positioner (ZDK) compared to subjects not using the ZDK. Patients electing to undergo primary TKA will be recruited into the study and randomized to receive and follow the ZDK protocol post-operatively or standard of care rehabilitation instructions. Knee extension measurements will be recorded at 2 weeks post-op and patient-reported outcome measurements will be recorded pre-operatively and at various post-op timepoints.

DETAILED DESCRIPTION:
Total Knee Arthroplasty (TKA) remains one of the most commonly performed elective surgical procedures in the United States. The number of TKAs performed annually has increased steadily since 2005 and is projected to be more than 3 million procedures annually by 2030. This steady growth may be attributed to the increasing geriatric population which is expected to represent 17% of the world's population by 2050. TKA aims to reduce pain and restore motion from those with knee complications, and with the geriatric population continuing to rise, TKA procedures are projected to grow over the next decade and beyond.

Historically, one of the major concerns following TKA is joint stiffness and subsequent range of motion loss. Range of motion loss, or more specifically, the inability to regain full extension (flexion contracture) have a relatively high occurrence and may lead to gait abnormalities and associated complications of the hips and low back. Early rehabilitation interventions following TKA may shorten the time needed to regain baseline extension/full extension and gait mechanics which not only is this beneficial for patient reported outcomes, but early rehabilitation interventions may reduce the economic burden associated with TKA recovery.

In-home or virtual physical therapy (PT) has also helped offload the economic burden to patients following TKA comparted to traditional in-clinic physical therapy. More importantly, the rise in in-home/virtual PT has not compromised patient outcomes, rather, it has improved them. In-home/virtual PT has reported improvements in total cost of therapy, compliance with unsupervised therapy, and hospital readmission rates.

Patient positioning has always played a vital role in the effectiveness of postoperative therapy. Historically, a continuous passive motion (CPM) machine was the standard for initiating ROM exercises, however, this modality has fallen out of favor due to the inconsistency of patient position and appropriate fitting of the device. The Zero Degree Knee (ZDK) positioning device is a knee extension pillow designed to simplify knee extension exercise following TKA surgery. Following knee surgery, the patient often experiences postoperative surgical pain which may lead to apprehension to physical therapy and engaging knee musculature. This apprehension may lead to joint stiffness and ultimately, ROM loss. The ZDK is a pillow that elevates the lower extremity and allows gravity to pull the knee passively and gently into an extended position. Additionally, the ZDK has a sliding capability that allows a patient to work on knee extension exercises along with knee flexion exercises.

In this study, the investigators aim to prospectively evaluate early post-operative knee extension and self-reported outcomes in patients using the Zero Degree Knee positioner. Patients electing to undergo primary TKA will be recruited into the study and randomized to receive and follow the ZDK protocol post-operatively or standard of care rehabilitation instructions. Knee extension measurements will be recorded at 2 weeks post-op and patient-reported outcome measurements will be recorded pre-operatively and at various post-op timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 40-80 years
* Candidate for total knee arthroplasty
* Diagnosis of mild to advanced osteoarthritis
* The ability to walk independently at baseline

Exclusion Criteria:

* History of knee replacement in operative limb (i.e. patients undergoing revision surgery)
* Neuromuscular/skeletal or connective tissue conditions that can alter gait or joint mechanics (joint infection, gout, rheumatoid arthritis)
* Pregnant women
* Prisoners
* Non-English speakers

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of the Zero Degree Knee device on post-operative knee extension in patients at 2 weeks post-op following total knee replacement as measured by lateral radiograph and physician interpretation. | 2 weeks
  The degree of knee extension at the 2 week post-operative visit will be measured via lateral radiograph interpreted by an orthopedic surgeon.

SECONDARY OUTCOMES:
Effect of the Zero Degree Knee device on PROMIS Physical Function scores in patients undergoing total knee replacement surgery. | 3 months
  Patient reported outcomes will be collected utilizing the Patient Reported Outcome Measurement Information Systems (PROMIS) Physical Function assessment tool. Patients receiving either the Zero Degree Knee device or standard of care rehabilitation instructions will complete PROMIS Physical Function assessment at the time of enrollment and at 2 weeks, 4 weeks, and 3 months after surgery. As the PROMIS tool has national normative data for age, sex, and condition, collection of patient-reported outcomes in this manner will allow for comparison between patients receiving the Zero Degree Knee device and standard of care as well as the general population. PROMIS Physical Function scores range from 0 to 100 and an increased PROMIS Physical Function score indicates an improvement in patient-reported physical function.
Effect of the Zero Degree Knee device on PROMIS Pain Interference scores in patients undergoing total knee replacement surgery. | 3 months
  Patient reported outcomes will be collected utilizing the Patient Reported Outcome Measurement Information Systems (PROMIS) Pain Interference assessment tool. Patients receiving either the Zero Degree Knee device or standard of care rehabilitation instructions will complete PROMIS Physical Function assessment at the time of enrollment and at 2 weeks, 4 weeks, and 3 months after surgery. As the PROMIS tool has national normative data for age, sex, and condition, collection of patient-reported outcomes in this manner will allow for comparison between patients receiving the Zero Degree Knee device and standard of care as well as the general population. PROMIS Pain Interference scores range from 0 to 100 and a decreased PROMIS Pain Interference score indicates an improvement in patient-reported pain interference.
Effect of the Zero Degree Knee device on PROMIS Mobility scores in patients undergoing total knee replacement surgery. | 3 months
  Patient reported outcomes will be collected utilizing the Patient Reported Outcome Measurement Information Systems (PROMIS) Mobility assessment tool. Patients receiving either the Zero Degree Knee device or standard of care rehabilitation instructions will complete PROMIS Physical Function assessment at the time of enrollment and at 2 weeks, 4 weeks, and 3 months after surgery. As the PROMIS tool has national normative data for age, sex, and condition, collection of patient-reported outcomes in this manner will allow for comparison between patients receiving the Zero Degree Knee device and standard of care as well as the general population. PROMIS Mobility scores range from 0 to 100 and an increased PROMIS Mobility score indicates an improvement in patient-reported mobility.
Effect of the Zero Degree Knee device on KOOS scores in patients undergoing total knee replacement surgery. | 3 months
  Patient reported outcomes will be collected utilizing the Knee Injury and Osteoarthritis Outcome Score (KOOS) tool. Patients receiving either the Zero Degree Knee device or standard of care rehabilitation instructions will complete the KOOS assessment at the time of enrollment and at 2 weeks, 4 weeks, and 3 months after surgery. The KOOS tool will allow for a comparison of scores of patients receiving the Zero Degree Knee device and standard of care. The maximum score a patient can achieve is 100, which indicates no knee problems. The minimum score a patient can achieve is zero, which indicates severe knee problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health - Midlands, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Result] Fortier LM, Rockov ZA, Chen AF, Rajaee SS. Activity Recommendations After Total Hip and Total Knee Arthroplasty. J Bone Joint Surg Am. 2021 Mar 3;103(5):446-455. doi: 10.2106/JBJS.20.00983. PMID 33337819
- [Result] Su EP. Fixed flexion deformity and total knee arthroplasty. J Bone Joint Surg Br. 2012 Nov;94(11 Suppl A):112-5. doi: 10.1302/0301-620X.94B11.30512. PMID 23118396
- [Result] Prvu Bettger J, Green CL, Holmes DN, Chokshi A, Mather RC 3rd, Hoch BT, de Leon AJ, Aluisio F, Seyler TM, Del Gaizo DJ, Chiavetta J, Webb L, Miller V, Smith JM, Peterson ED. Effects of Virtual Exercise Rehabilitation In-Home Therapy Compared with Traditional Care After Total Knee Arthroplasty: VERITAS, a Randomized Controlled Trial. J Bone Joint Surg Am. 2020 Jan 15;102(2):101-109. doi: 10.2106/JBJS.19.00695. PMID 31743238
- [Result] Harvey LA, Brosseau L, Herbert RD. Continuous passive motion following total knee arthroplasty in people with arthritis. Cochrane Database Syst Rev. 2014 Feb 6;2014(2):CD004260. doi: 10.1002/14651858.CD004260.pub3. PMID 24500904